CLINICAL TRIAL: NCT06926335
Title: Oncological Safety of Oncoplastic Breast Surgery in Multicentric Breast Retrospective Study
Brief Title: Oncological Safety of Oncoplastic Breast Surgery in Multicentric Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshymaa Abd-Elhars Ebrahem, General Surgery Resident, Assiut University
Other Study IDs: Breast conserve
Record Dates: First submitted 2025-04-01; First posted 2025-04-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Safety of Breast Coservative Multicenteric Breast Cancer; Breast Neoplasms; Breast Cancer; Multicentric
Keywords: Breast conservative surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: Breast consevative surgery — plastic surgery principles within the context of sound oncological resection. Volume-reducing or volume- replacing methods are utilised to optimise postoperative appearances whilst prioritizing negative margin resection, supported by prompt adjuvant therapy

SUMMARY:
The purpose of the study is to evaluate Oncological safety of oncoplastic breast surgery in multicentric breast cancer

DETAILED DESCRIPTION:
Breast cancer is the most prevalent cancer in women worldwide, accounting for about 23.8%. Multifocal and multicentric breast tumors are defined as two or more neoplasms separated in one breast. In multifocal tumors, a quarter of the breast is involved while in multicentric tumors, two quarters or more are involved. There is no exact radiological definition, but the distance between the multifocal tumors is less than or equal to 5 cm, whereas the distance between multicentric tumors is 5 cm, or more.

Due to increasingly use of more developed imaging methods such as tomosynthesis, magnetic resonance imaging (MRI) in these patients, we face more MF/MC breast cancer cases. It is seen that MF/MC breast cancer incidence ranges from 6% to 75% in different series.

Breast-conserving surgery (BCS) and radiotherapy have been adopted as the main treatment methods for early breast cancer. However, there are some studies stating that BCS carries risks for local recurrence in patients with MF/MC breast cancer.

Oncoplastic breast conservation (OBC) relies on applying plastic surgery principles within the context of sound oncological resection. Volume-reducing or volume- replacing methods are utilised to optimise postoperative appearances whilst prioritizing negative margin resection, supported by prompt adjuvant therapy. In fact, it is agreed that in cases where more than 20% of the breast tissue must be excised for oncological margin clearance, oncoplastic surgery is likely to require more complex techniques.This may allow larger specimens to be resected than in traditional breast conservation surgery, but with comparable histopathological properties to those who would be offered mastectomy.

Previous work has suggested that as such, OBC should be regarded as a separate entity from breast conservation therapy, and that direct comparison with mastectomy outcomes should be performed to inform decision-making amongst clinicians and with patients when planning for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with multicentric breast cancer
* Female Patient aged from 18 to 65 years old
* Patients who are fit for general anesthesia.
* Patients who provide a written informed consent.
* Patient who agree to provide short term outcome data and agree to provide contact information to provide contact information

Exclusion Criteria:

* Female patients less than 20 years old
* Stage 4 breast cancer
* Patients who are contraindicated for radiotherapy
* Pregnant patients in first trimester
* Patient with inflammatory carcinoma

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients of multicentric breast cancer underwent oncoplastic breast surgery from 2020 to 2025
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
To evaluate Oncological safety of oncoplastic breast surgery in multicentric breast cancer | 5 years
  Number of multicentric breast cancer who underwent breast conservative surgery with no recurrance

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Egypt